CLINICAL TRIAL: NCT03772028
Title: Phase III Randomized Clinical Trial for Stage III Epithelial Ovarian Cancer Randomizing Between Primary Cytoreductive Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Primary Cytoreductive Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Acronym: OVHIPEC-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M17OVH; ENGOT-ov52/DGOG/OVHIPEC-2 (Other: European Network of Gynaecological Oncological trials Groups)
Record Dates: First submitted 2018-09-21; First posted 2018-12-11 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; HIPEC; OVHIPEC; primary debulking
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: randomized controlled, open-label, multicenter phase III trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- conventional surgery (No Intervention): Primary cytoreductive surgery without HIPEC
- HIPEC (Experimental): Primary cytoreductive surgery with HIPEC with cisplatin
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: cisplatin — HIPEC with cisplatin after cytoreductive surgery
  Arms: HIPEC

SUMMARY:
stage III epithelial ovarian cancer randomizing between primary cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy

DETAILED DESCRIPTION:
The objective of this study is to prove that treatment with primary cytoreductive surgery in combination with HIPEC (treatment arm) improves outcome compared to primary cytoreductive surgery without HIPEC (standard arm) with acceptable morbidity, in patients with FIGO stage III epithelial ovarian cancer who are eligible for primary cytoreductive surgery with no residual disease, or residual disease up to 2.5 mm.

ELIGIBILITY:
Inclusion Criteria:

* candidate for primary CRS
* histological or cytological proven FIGO stage III primary epithelial ovarian, fallopian tube, or extra-ovarian cancer

Exclusion Criteria:

* history of previous malignancies within 5 years prior to inclusion
* FIGO stage IV disease
* complete primary cytoreduction is impossible
* prior treatment for the current malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ovarian cancer
Enrollment: 538 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year after last patient last visit

SECONDARY OUTCOMES:
recurrence-free survival | 1 year after last patient last visit
adverse events | 30 days after end of treatment
  toxicity of extra treatment compared standaard treatment
cost evaluation | 1 year after lplv
  cost evaluation based measured by quality adjusted life year

CONTACTS AND LOCATIONS:
Locations (28):
- United States (2):
  - City of Hope, Duarte, California
  - MSKCC New York, New York, New York
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- France (11):
  - CHU de Besancon, Besançon
  - Institut Bergonié, Bordeaux
  - o Institut Bergonié, Bordeaux, Bordeaux
  - CHU Lille, Lille
  - Centre Leon Berard, Lyon, Lyon
  - CHU Lyon, Lyon
  - Institut du Cancer Montpellier, Montpellier
  - Institut de Cancerologie de l'Ouest, ICO Nantes), Nantes
  - Institut Curie Paris, Paris
  - CHRU Strasbourg, Strasbourg
  - Oncopole, Institute Universitaire du Cancer de Toulouse (IUCT Toulouse), Toulouse
- Mater Misericordiae University Hospital, Dublin, Dublin, Ireland
- Italy (2):
  - Policlinico Sant'Orsola, Bologna, Bologna
  - Fondazione Policlinico A Gemelli IRCCS, Roma
- Netherlands (10):
  - Antoni van leeuwenhoek, Amsterdam, North Holland
  - Amsterdam UMC, Amsterdam
  - Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - UMCG, Groningen
  - Leiden University Medical Center (LUMC), Leiden
  - Maastricht UMC+, Maastricht
  - Radboud MC, Nijmegen
  - Erasmus MC, Rotterdam
  - UMCU, Utrecht
- Alice Bjoernlund-Larsen, Uppsala, Sweden

REFERENCES:
- [Derived] Koole S, van Stein R, Sikorska K, Barton D, Perrin L, Brennan D, Zivanovic O, Mosgaard BJ, Fagotti A, Colombo PE, Sonke G, Driel WJV; OVHIPEC-2 Steering Committee and the Dutch OVHIPEC group. Primary cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy (HIPEC) for FIGO stage III epithelial ovarian cancer: OVHIPEC-2, a phase III randomized clinical trial. Int J Gynecol Cancer. 2020 Jun;30(6):888-892. doi: 10.1136/ijgc-2020-001231. Epub 2020 Mar 23. PMID 32205449